CLINICAL TRIAL: NCT06026774
Title: A Clinical Study to Assess the Safety, Feasibility, and Efficacy of Personalized mRNA Vaccine Encoding Neoantigen in Combination With Standard Adjuvant Therapy in Subjects With Resected Digestive System Neoplasms
Brief Title: Clinical Study of Personalized mRNA Vaccine Encoding Neoantigen in Subjects With Resected Digestive System Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiujun Cai, The director of Sir Run Run Shaw Hospital, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2023-755-03
Record Dates: First submitted 2023-08-25; First posted 2023-09-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Digestive System Neoplasms
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNeo-Vac-R01 in combination with standard adjuvant therapy (Experimental): Subjects will receive at least 4 cycles of standard adjuvant therapy according to CSCO clinical guidelines after surgery. Then subjects will receive iNeo-Vac-R01 via IH injection on Day 1 of each 21-day cycle for up to 9 cycles at an applicable dose, identified during the dose escalation phase of the study.
  Interventions: Biological: iNeo-Vac-R01 in combination with standard adjuvant therapy

INTERVENTIONS:
Biological: iNeo-Vac-R01 in combination with standard adjuvant therapy — Personalized mRNA vaccine encoding neoantigen, IH injection

SUMMARY:
The purpose of this study is to assess the safety, feasibility, and efficacy of personalized mRNA vaccine iNeo-Vac-R01 with standard adjuvant therapy in subjects with surgically resected digestive system neoplasms.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm clinical study of personalized mRNA vaccine iNeo-Vac-R01 in combination with standard adjuvant therapy in subjects with surgically resected digestive system neoplasms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >/= 18 years old and </= 75 years old, with the ability to understand and provide signed and witnessed informed consent, and agree and are able to comply with protocol requirements.
2. Subjects must have one of the histologically- or cytologically-confirmed advanced (locally advanced or metastatic) digestive system neoplasms listed below that can be radical resected. Subjects must be able to receive at least 4 cycles of standard adjuvant therapy according to CSCO clinical guidelines after surgery. The toxic effects of previous anti-tumor treatments have returned to </= grade 1 defined by NCI-CTCAE v5.0 or to the level specified by the inclusion/exclusion criteria.

   Subjects with any of the following digestive system neoplasms:

   a. Cholangiocarcinoma b. Pancreatic cancer c. Hepatocellular carcinoma d. Gastric cancer e. Colorectal carcinoma
3. Expected survival >/= 6 months.
4. ECOG performance status score of 0 ~ 1.
5. Sufficient tumor tissue samples can be obtained from subjects for genetic analysis, with at least 0.5cm*0.5cm of tissue required for surgical samples.
6. Echocardiographic evaluation: left ventricular ejection fraction (LVEF) >/= 50%.
7. The organ function level must meet the following requirements: absolute neutrophil count (ANC) >/= 1.5 × 10^9/L, platelet count (PLT) >/= 80 × 10^9/L, hemoglobin (Hb) >/= 90 g/L; serum total bilirubin (TBIL) </= 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 × ULN (if there is liver metastasis, TBIL </= 3 × ULN, AST, ALT </= 5 ×ULN are allowed), serum albumin >/= 28g/L, serum creatinine </= 1.5 × BUN, Glomerular filtration rate >/= 50mL/min, prothrombin time (PT) and activated partial thromboplastin time (APTT) and international standardized ratio (INR) </= 1.5 × ULN (without anticoagulant therapy) .
8. For women of childbearing potential: having a negative serum or urine pregnancy test within 7 days prior to study initiation, agreement to remain abstinent or use contraceptive measures during the treatment period.
9. For men: agreement to remain abstinent or use contraceptive measures during the treatment period.

Exclusion Criteria:

1. Subjects with cancer requiring anti-tumor treatment within the 5 years prior to enrollment in the study (except stage I prostate cancer, cervical cancer in situ, breast cancer in situ, papillary thyroid cancer and non-melanoma skin cancer that have been treated).
2. Subjects who received major surgery, or had obvious traumatic injury or long-term untreated wounds or fractures within 2 weeks prior to the first dose of iNeo-Vac-R01.
3. Subjects whose sequencing data was found that there are no new antigens available for individualized immunotherapy after analysis.
4. Subjects who prepare to undergo or have previously received bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation. Subjects who receive other anti-tumor treatments within 2 weeks prior to the first dose of iNeo-Vac-R01, including surgical treatment, chemotherapy, radiation therapy, targeted therapy, endocrine therapy, immunotherapy, biological therapy, interventional therapy, or other clinical trial related treatments.
5. Subjects who need to use immunosuppressants, or systemic or absorbable local glucocorticoids therapy to achieve immunosuppressive effects and continue to use them within 7 days before the first administration (excluding those with daily doses of glucocorticoids less than 10mg of prednisone or doses of other therapeutic glucocorticoids equal to 10mg of prednisone).
6. Subjects who received other vaccines within 4 weeks before the first dose of iNeo-Vac-R01, and are expected to receive other vaccines during treatment period of the study or within 60 days after the last dose of iNeo-Vac-R01.
7. Subjects who have an active infection or uncontrollable infection requiring systemic treatment, including fungi, bacteria, viruses, or other infections; subjects with active tuberculosis;
8. Subjects with positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb) and positive hepatitis B virus DNA titer detection greater than normal range; positive hepatitis C virus (HCV) antibody and HCV RNA detection greater than normal range; positive human immunodeficiency virus antibody; positive treponema pallidum-specific antibody.
9. Subjects with autoimmune diseases or immune deficiencies treated with immunosuppressive drugs, except vitiligo, type 1 diabetes, autoimmune hypothyroidism requiring hormone treatment and psoriasis not requiring systemic treatment; known history of primary immunodeficiency.
10. Subjects with cardiocerebrovascular events: previously or currently heart valve disease >/= grade 3, heart failure within 8 weeks before the first dose of iNeo-Vac-R01 (New York Heart Association [NYHA] cardiac function >/= grade II, myocardial infarction, unstable angina, stroke, transient ischemic attack, cardiac surgery (including coronary artery bypass grafting or percutaneous coronary intervention) within 8 weeks before the first dose of iNeo-Vac-R01, concomitant severe electrocardiogram abnormalities (such as ventricular flutter, ventricular fibrillation, multiform ventricular tachycardia, sick sinus syndrome, third degree atrioventricular block without pacemaker treatment, QTc >/= 480ms, and other conditions evaluated by the investigators as severe abnormalities), hypertension with poor drug control (systolic blood pressure >/= 160mmHg and/or diastolic blood pressure >/= 100mmHg), or other cardiocerebrovascular diseases that have been evaluated by the investigators as unsuitable for participation in this trial.
11. Subjects with respiratory disease: previously or currently pulmonary fibrosis, interstitial lung disease, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe asthma, pulmonary hypertension or severe impairment of lung function, etc.
12. Subjects with moderate to severe ascites with clinical symptoms; uncontrolled or moderate to equal amounts of pleural effusion and pericardial effusion.
13. Subjects with drug abuse; clinical or psychological or social factors that affect informed consent or research implementation.
14. Subjects with a history of allergies to immunotherapy or vaccines, or other potential immunotherapy allergies identified by the investigators.
15. Subjects identified that it is not suitable for enrollment or may not be able to complete this experiment for other reasons by the investigators.
16. Vulnerable groups, including individuals with mental illness, cognitive impairment, critical patients, minors, pregnant or lactating women, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-08 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) [safety and tolerability] | 21 days after last iNeo-Vac-R01 dose

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years after first dose of iNeo-Vac-R01
  OS is defined as time between the date of the first dose of iNeo-Vac-R01 and the date of death due to any cause.
Recurrence Free Survival (RFS) | 3 years after first dose of iNeo-Vac-R01
  RFS is defined as time between the date of first dose of iNeo-Vac-R01 and the date of either disease recurrence or death (whichever is sooner).
The proportion of subjects who have no disease recurrence at 12 months or 24 months after first dose of iNeo-Vac-R01. | 12 months and 24 months after first dose of iNeo-Vac-R01
Neoantigen-specific T Cell Response [immunogenicity] | 12 months after first dose of iNeo-Vac-R01
  Detect the level of specific TNF-γ in peripheral blood of subjects by ELISpot in order to measure the neoantigen-specific T cell response of subjects.
T Cell Subsets [immunogenicity] | 12 months after first dose of iNeo-Vac-R01
  Detect the proportion of different T cell subsets in T cells by flow cytometry.
Cytokines Level [immunogenicity] | 6 months after first dose of iNeo-Vac-R01
  Record the changes of IL-2, IL-6, IL-8, IL-10, IL-12, and TNF-α in peripheral blood before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China